CLINICAL TRIAL: NCT01044810
Title: Comparison of Virological and Immunological Results of Efavirenz-based Regimen in HIV-infected Patients With or Without Allergic Reactions to Nevirapine
Brief Title: Effectiveness of Efavirenz-based Regimen in HIV-1-infected Patients With Nevirapine Hypersensitivity
Status: Completed | Type: Observational
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Collaborators: Thai Red Cross AIDS Research Centre (Other); Clinical Research Collaborative Network (Network)
Responsible Party: Krittaecho Siripassorn, Bamrasnaradura Infectious Diseases Institute
Other Study IDs: BIDI-EFV
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Treatment Failure, HIV or AIDS; CD4 Cell Counts
Keywords: HIV; efavirenz; nevirapine; allergy; rash; Cohort Studies, Historical; Retrospective Study; exanthem; Antiretroviral Agents; Highly Active Antiretroviral Therapy; HAART; treatment failure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypersensitivity; Exanthema | interventions — efavirenz

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Simultaneous interruption (Exposure gr): stopped all drugs in NNRTI-based regimens simultaneously after allergic reactions to NVP-based regimens, and later started EFV-based regimens
  Interventions: Drug: Efavirenz-based regimens
- Naive (Control group): HIV-1-infected patients who started EFV-based regimens as their initial ARV regimens.
  Interventions: Drug: Efavirenz-based regimens
- staggered interruption (exposure group): after having allergic reactions to NVP-based regimens, stopped NNRTIs first, continued the other NRTIs for a period of time, i.e. "staggered interruption", and later started EFV-based regimens
  Interventions: Drug: Efavirenz-based regimens

INTERVENTIONS:
Drug: Efavirenz-based regimens — Efavienz: 600 mg, oral, every 24 hours, continued medication until the end of study.
  Other Names: Stocrin, Sustiva

SUMMARY:
The primary objective of this study is to compare the effectiveness of EFV-based regimens in HIV-1-infected patients who; (1) were previously allergic to NVP and stopped all ARV simultaneously; (2) were previously allergic to NVP and continued the other NRTIs for a period of time, i.e. "staggered interruption"; and (3) started EFV-based regimens as an initial regimen (as controlled group).

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years old
* documented HIV infection
* started EFV-based regimens between January 2002 and December 2008 at Bamrasnaradura Infectious Diseases Institute

Exclusion Criteria:

* previously received non-HAART regimens such as dual NRTIs regimen, AZT monotherapy with single-dose NVP in pregnancy patients
* previously received protease inhibitor-based regimen
* diseases or conditions that significantly affected either kidney or liver functions such as decompensated liver cirrhosis, ESRD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who started EFV-based regimens between January 2002 and December 2008 at Bamrasnaradura Infectious Diseases Institute
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time to Virological failure | until end of study cohort
  Virological failure was defined as either (1) two consecutive results of plasma HIV-1 RNA >400 copies/ml or (2) plasma HIV-1 RNA >1,000 copies/ml with genotypic resistance assay revealed NRTI or NNRTI resistance-associated mutations

SECONDARY OUTCOMES:
Virological suppression | 24 months
  Virological suppression was defined as having plasma HIV-1 RNA <50 copies/ml
Median increase from baseline of CD4 cell count | 24 months
Adverse events | until end of cohort
  Adverse events were defined as either (1) having more than grade 3 according to DAID AE Grading Table, or (2) having clinical events that leaded to changed antiretroviral medications
Clinical outcomes such as death, major opportunistic infections, immune recovery syndrome, non-AIDS events | until end of cohort

CONTACTS AND LOCATIONS:
Overall Officials: Krittaecho Siripassorn, MD, Principal Investigator — Bamrasnaradura Infectious Diseases Institute
Locations (1):
- Bamrasnaradura Infectious Disease Institute, Nonthaburi, Thailand